CLINICAL TRIAL: NCT00893503
Title: Stop Colorectal Cancer Through Prevention and Screening
Brief Title: Scope Pilot Research Study
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other)
Responsible Party: Dr. Daniel C. Sadowski, Royal Alexandra Hospital
Other Study IDs: AHS-160408-SP; Pro00002130
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: colonoscopy — Patients will provide stool and urine samples and will be scheduled to undergo a colonoscopy. The colonoscopy will be done per standard of care - no study specific procedural requirements imposed.
  Other Names: Endoscopy

SUMMARY:
Colorectal cancer is a major public health concern in Alberta. Colorectal Cancer is the fourth most common diagnosed cancer and second overall in terms of cancer deaths in Canada. One in 14 males and 1 in 16 females aged 50-74 will be diagnosed with colorectal cancer and will have an overall 1 in 28 chance of dying from colorectal cancer. While colorectal cancer is surgically curable if diagnosed in the early stages, with five year survival rates of 90% versus 10% if detected at more advanced stages, less than 20 % of all individuals in this age bracket traditionally have undergone colorectal cancer screening. Colorectal cancer often presents with non-specific symptoms where non-cancerous polyps are commonly found. If these polyps are left in place, they may grow over time and progress from a non-cancerous mass to symptomatic cancerous tumors; therefore, early screening in those patients without symptoms may thereby prevent the progression from a non-cancerous to cancerous finding.

The hypothesis, or theory being studied in the SCOPE Pilot research study, is that implementation of a colorectal screening program would decrease colorectal cancer prevalence, increase the long-term survival ratio for patients, and decrease burden on the health care system. Moreover, early detection and treatment of colorectal cancer has the potential to increase the lifespan of patients and decrease health care costs.

The SCOPE Pilot Research study will recruit 1000 individuals between the ages of 50 - 74 of average to high risk for developing colorectal cancer as determined by their referring Gastroenterologists. Those patients who are ages 40-50 will also be eligible if they have a personal or family history of colorectal cancer. Patients referred to the SCOPE Pilot program will be further screened for eligibility, and if no exclusion criterion is present, will be invited to attend an education session and research program. The SCOPE Pilot research study will compare the current fecal occult blood testing (FOBT - Hemoccult II) with newly available FOBT blood testing along with colonoscopy therapy. It will also encompass educational information, risk stratification, screening for both average and high risk patients, and colonoscopy.

DETAILED DESCRIPTION:
In the Capital Health Region, 18.6% of colorectal cancers are detected at stage 1, while 22.4% are already at stage IV. The Capital Health Region has 340,000 individuals aged 50-74, yet only 14.3% receive any colorectal cancer screening. These low screening rates may be attributed to lack of awareness, the limitations of the fecal occult blood testing (FOBT) and the unpleasant associations with both the FOBT and the colonoscopy. The limitations of the FOBT include low sensitivity for detection of adenomas and small cancers, the cumbersome method of stool collection on multiple days and the dietary restrictions, which make patient compliance low and introduce high probability of false positive tests and unnecessary colonoscopies.

Currently, there are two screening modalities available. The fecal occult blood testing (FOBT: Hemoccult II) detects blood in the stool that may be due to colonic adenomas or cancer. The second is colonoscopy, which is the gold standard in detecting colorectal lesions; however it carries the risks of bleeding and bowel perforation. FOBT is the recommended primary screening tool for patients at average risk for developing colorectal cancer. Large population-based randomized controlled trials have consistently demonstrated a significant survival benefit in patients who undergo annual or biannual screening with FOBT.

Recently, newer generation FOBT techniques, the FOBT immunochemical (FIT) has become available. These tests are more sensitive in detecting specifically human blood in the stool and do not require dietary restrictions. Recent studies have suggested the diagnostic performance of the FIT may be superior to standard Hemoccult II rates because of simplified sampling. As well, economic analysis have suggest that the use of FIT is superior to FOBT in diagnostic performance at a reasonable cost to a European population.

A urine specimen will also be obtained and analyzed for metabolomics for each subject. Metabolomics is the study of the global chemical composition of an organism. It utilizes technologies such as a nuclear magnetic resonance spectroscopy to study the metabolite / chemical composition, interactions, and changes in these levels in response to disease or environmental factors. By analyzing urine samples, it has been possible to identify the metabolite patterns characteristic of various diseases. In addition, the metabolite patterns of liver disease caused by cirrhosis and hepatitis, inflammatory bowel disease and cancer have been identified. Urine metabolomics analysis may offer a new sensitive, yet inexpensive screening tool for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients on gastrointestinal wait-lists for screening colonoscopy
* patients that are 50 - 75 years of age at average risk for colorectal cancer OR patients that are 40 - 75 years of age and at high risk for colorectal cancer
* Patients that are healthy or have co-morbidities that are currently stable
* patients that are willing to complete 1 FOBT, 2 FITs, urine for metabolomics, attend an education session, colonoscopy and evaluate the SCOPE program and education resources.
* individuals will be eligible to participate in the pilot if their last colonoscopy was a minimum of five (5) years ago. Less than 5 years is acceptable if the procedure report on the last colonoscopy recommends repeat colonoscopy at an earlier interval.

Exclusion Criteria:

* under 40 years of age or over 75 years of age
* inability to understand / sign informed consent (applies to individuals that do not speak or read English)
* use of warfarin or any anticoagulant medications (includes low molecular weight heparin)
* rectal bleeding
* past history of failed or extremely difficult colonoscopy
* insulin dependent diabetes
* history of inflammatory bowel disease
* use of Bi-pap or home oxygen
* Asthma or COPD described as severe
* chronic disease that is suspected / under investigation but NYD
* chronic / acute disease process that is not stable or not in remission
* possible lynch syndrome
* renal disease requiring any type of dialysis
* BMI > 35

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Family practitoners will refer patients to Gastroenterologist physicians for consideration into the SCOPE Pilot Research program. They will be evaluated for suitability initially by gastroenterologists who will then refer them directly to the SCOPE Pilot research program to further assess suitability. Those patients who meet the inclusion criteria with no exclusion criteria present will be invited to an education session and invited to partake in the research program if willing.
Sampling Method: Non-Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic performance characteristics of the guaiac based Hemoccult II FOBT and two FIT's, the Hemoccult ICT and MagStream HemSp, using colonoscopy as the gold standard. | FOBT, FIT (Hemoccult ICT) and MagStream Hemsp will be obtained prior to colonoscopy.

SECONDARY OUTCOMES:
Estimate the probability of participants of the SCOPE pilot who have adenomas or colorectal cancer using urine metabolomics and correlate those with results from the FOBT / FIT's and screening colonoscopy. | Urine sample obtained prior to colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Sadowski, MD, Principal Investigator — Royal Alexandra Hospital; Richard N Fedorak, MD, Study Director — University of Alberta; Clarence K Wong, MD, Study Director — Royal Alexandra Hospital
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Walter C. MacKenzie Centre, University of Alberta, Edmonton, Alberta